CLINICAL TRIAL: NCT03975764
Title: Fecal Microbiota in Preterm Birth
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ola Gutzeit MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0120-18
Record Dates: First submitted 2019-06-02; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Gut Microbiome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal semple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm birth: Delivery between 24-32 weeks of gestation
  Interventions: Diagnostic Test: Collection of fecal sample
- Term delivery: Delivery between 37-41 weeks of gastation
  Interventions: Diagnostic Test: Collection of fecal sample

INTERVENTIONS:
Diagnostic Test: Collection of fecal sample — Analysis of fecal microbiome

SUMMARY:
We will compeer fecal microbiome in preterm birth with fecal microbiome of team labor

ELIGIBILITY:
Inclusion Criteria:

* Woman after vaginal delivery of singleton

Exclusion Criteria:

* Fetal abnormalities
* Gestational diabetes
* Hypertensive disorder

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Woman after vaginal delivery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Unique microbial fingerprint | 1 year
  16S rRNA gene sequencing

IPD SHARING:
Plan to Share IPD: No